CLINICAL TRIAL: NCT00350272
Title: A Randomized, Blinded, 12-week Comparison of Elvucitabine/Efavirenz/Tenofovir Versus Lamivudine/Efavirenz/Tenofovir in HIV-1 Infected Treatment-naive Participants. There is a 36 Week, Open-label, Extension Phase for Eligible Participants.
Brief Title: Elvucitabine/Efavirenz/Tenofovir Versus Lamivudine/Efavirenz/Tenofovir in Human Immunodeficiency Virus (HIV)-1 Infected, Treatment-naive Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH443-015
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: HIV-1 treatment naive
MeSH Terms: conditions — HIV Infections | interventions — dexelvucitabine; Lamivudine; Tenofovir; efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elvucitabine, Efavirenz, Tenofovir (Experimental): Elvucitabine (blinded) 10 milligrams (mg)/day in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
  Participants who experienced at least a 2 log10 decrease in HIV-1 RNA from Baseline or who had an HIV-1 RNA level of less than 400 copies/ mL at Week 10 and had not experienced any Grade 3 or 4 hematological toxicity as of the Week 10 measurement were considered eligible for an additional 84 weeks of open-label treatment after Week 12.
  Interventions: Drug: Elvucitabine; Drug: Tenofovir; Drug: Efavirenz
- Lamivudine, Efavirenz, Tenofovir (Active Comparator): Lamivudine (blinded) 300 mg daily in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
  Participants who experienced at least a 2 log10 decrease in HIV-1 RNA from Baseline or who had an HIV-1 RNA level of less than 400 copies/mL at Week 10 and had not experienced any Grade 3 or 4 hematological toxicity as of the Week 10 measurement were considered eligible for an additional 84 weeks of open-label treatment after Week 12.
  Interventions: Drug: Lamivudine; Drug: Tenofovir; Drug: Efavirenz

INTERVENTIONS:
Drug: Elvucitabine — Elvucitabine 10 mg orally daily
  Other Names: ACH-126,443
  Arms: Elvucitabine, Efavirenz, Tenofovir
Drug: Lamivudine — Lamivudine 300 mg orally daily
  Other Names: 3TC
  Arms: Lamivudine, Efavirenz, Tenofovir
Drug: Tenofovir — Tenofovir open-label 300 mg orally daily
  Other Names: Viread
Drug: Efavirenz — Efavirenze open-label 600 mg orally daily
  Other Names: Sustiva

SUMMARY:
Elvucitabine, a novel nucleoside analog, is being studied as a treatment for participants with human immunodeficiency virus (HIV)-1. This Phase 2 study will enroll 60 HIV-1-naive participants to assess the efficacy and safety of elvucitabine compared to lamivudine in combination with tenofovir and efavirenz as measured by changes in the participant's HIV-ribonucleic acid (RNA) level and CD4 cell count. The study treatment will be 12 weeks of blinded study medication followed by an additional 84 weeks of open-label treatment if the participant's response to treatment meets certain endpoints. The pharmacokinetics of elvucitabine will also be assessed during the study.

DETAILED DESCRIPTION:
Sixty HIV-1-infected, clinically stable, treatment-naïve adults with no acquired immunodeficiency syndrome (AIDS)-defining events during the 3 months prior to screening will be randomly assigned to 1 of 2 treatment groups. Participant plasma HIV-1 RNA levels must be greater than or equal to 5000 copies/millimeter (mL), and CD4 cell counts must be greater than 200 cells/mL and less than 500 cells/mL at Screening. Participants must be sensitive to elvucitabine, lamivudine, and emtricitabine as demonstrated by the absence of the M184V, M184I, and D237E mutations by TRUGENE HIV-1 Genotyping Kit. Participants must be genotypically sensitive to efavirenz (negative for K103 or Y188L mutations) and tenofovir (negative for K65R mutation) as demonstrated by TRUGENE HIV-1 Genotyping Kit. They must have acceptable hematologic and chemistry parameters.

Participants whose HIV-1 RNA levels have decreased at least 2 logs or to below 400 copies/mL by Week 10 may be considered eligible to enter the extension phase of up to 36 weeks of additional treatment. Participants in the extension phase will be evaluated at Weeks 14 and 16 and every 4 Weeks until Week 96.

Once all participants have completed 12 weeks of treatment, and the data are available for all visits through Week 12, the database will be locked and the treatment assignments will be unblinded. Any participant who has had less than 48 weeks of treatment will be allowed to continue on the same treatment as initially assigned on an open-label basis through 48 weeks. All participants will have 2 post-treatment follow-up visits, at 1 and 4 weeks after the end of treatment. Concentrations of elvucitabine in the plasma will be measured on Day 1, at Weeks 4, 6, 8, 12, 16, 24, 48, 72, 96, and at Follow-up

Efficacy will be assessed by measuring plasma HIV-1 RNA levels and CD4 counts at each study visit.

Safety evaluation will include vital signs, physical examinations, electrocardiograms, assessments of adverse events (AEs), measurement of plasma HIV-1 RNA levels and CD4 counts, determination of HIV-1 genotype at Screening and at Weeks 12, 24, 48, and 96, determination of HIV-1 phenotype at Visit 1 and at Weeks 12, 24, 48, and 96 urine and serum pregnancy tests, as well as laboratory analyses that include hematology, chemistry, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet the following criteria at Screening to be enrolled in this study:

1. Are male or female. Sexually active men with partners of childbearing potential must agree to use an acceptable form of contraception as determined by the investigator (for example, oral contraceptives, double-barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or vasectomy) during participation in the study. Female participants cannot be pregnant or lactating/breast-feeding and must be surgically sterile, postmenopausal as defined later, or practicing an effective method of birth control as determined by the investigator (for example oral contraceptives, double-barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy). A woman may be considered postmenopausal if she is at least 50 years or older, has a history of no menses for at least 12 months, and has a follicle-stimulating hormone (FSH) level over the upper limit of normal for reproductive aged women.
2. Are 18 through 65 years old
3. Have documented HIV-1 infection by written prior history and clinically stable with no AIDS-defining events in the 3 months prior to Screening
4. Have plasma HIV-1 RNA levels greater than or equal to 5000 copies/mL at Screening
5. Are HIV-1 strain sensitive to elvucitabine, lamivudine, or emtricitabine as demonstrated by the absence of the M184V, M184I, and D237E mutations by TRUGENE HIV-1 Genotyping Kit
6. Are HIV-1 strain genotypically sensitive to efavirenz (negative for K103 and Y188L mutations) and tenofovir (negative for K65R mutation) by TRUGENE HIV-1 Genotyping Kit
7. Have a CD4 count greater than or equal to 200 cells/mL and less than 500 cells/mL
8. Have acceptable hematologic and chemistry parameters, including the following:

   * Hemoglobin (Hgb) greater than or equal to 11 grams (g)/deciliter (dL)
   * Absolute neutrophil count greater than or equal to 2000 cells/mm^3
   * Platelets greater than or equal to 125 000/mm^3
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 1.5 times the upper limit of normal
   * Total bilirubin less than or equal to 1.5 times the upper limit of normal
   * Creatinine within normal range
9. Are capable of understanding and has signed the informed consent document
10. Are able and willing to comply with protocol requirements

Exclusion Criteria:

Participants meeting any of the following criteria at Screening will be excluded from the study:

1. Are hepatitis B surface antigen positive, and/or hepatitis B virus (HBV) deoxyribonucleic acid (DNA) positive
2. Have previous therapy with agents with significant systemic myelosuppressive or cytotoxic potential within the 3 months prior to Screening or the expected need for such therapy during the study
3. Have previous use or need for bone marrow colony-stimulating factors such as Epogen, Procrit, or Neupogen
4. Have had previous antiretroviral therapy
5. Have evidence or history of cirrhosis
6. Have recent (within 3 months of Screening) history of alcohol abuse, physical dependence to any opioid, cocaine, lysergic acid diethylamide (LSD) or amphetamines, or history of drug addiction within the last 12 months
7. Have inability to tolerate oral medication
8. Are pregnant or breast-feeding if female
9. Have any clinical condition or prior therapy that, in the investigator's opinion, would make the participant unsuitable for the study or unable to comply with the dosing requirements
10. Have received treatment with any other investigational drug within 30 days prior to Screening
11. Have current active mental illness or a history of significant mental illness (for example, severe depression, schizophrenia, history of suicidal ideations, or suicide attempts)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (20):
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, Long Beach, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Fort Myers, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Wichita, Kansas
  - Clinical Trial Site, Washington D.C, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Newark, New Jersey
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Hampton, Virginia
- Clinical Trial Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available to only this study's Principal Investigator upon request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Human immunodeficiency virus (HIV)-1-infected, treatment-naïve adults with no acquired immunodeficiency syndrome (AIDS)-defining events in the 3 months prior to Screening and with plasma HIV-1 ribonucleic acid (RNA) levels greater than or equal to 5000 copies/milliliter (mL) and CD4 counts greater than or equal to 200 cells/microliter (μL) and less than 500 cells/μL, and HIV-1 strains absent of the M184V, M184I, D237E, K103, Y188L, and K65R mutations at Screening.
Pre-assignment Details: A total of 78 participants were given a treatment assignment. One participant assigned to treatment was ineligible for randomization and did not receive any study drug. An additional participant did not take any of the dispensed study drug. Therefore, 76 participants were treated.
Groups:
- Elvucitabine, Efavirenz, Tenofovir: Elvucitabine (blinded) 10 milligrams (mg)/day in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
- Lamivudine, Efavirenz, Tenofovir: Lamivudine (blinded) 300 mg daily in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
Period: Blinded 12-Week Treatment
Arm/Group | Elvucitabine, Efavirenz, Tenofovir | Lamivudine, Efavirenz, Tenofovir
Started | 39 | 37
Completed | 30 | 35
Not Completed | 9 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Sponsor decision | 0 | 1
Period: Open-Label 84 Week Treatment
Arm/Group | Elvucitabine, Efavirenz, Tenofovir | Lamivudine, Efavirenz, Tenofovir
Started | 30 | 35
Completed | 21 | 27
Not Completed | 9 | 8
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Sponsor decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was the safety population, defined as all randomized participants who received at least one dose of the study drug.
Groups:
- Elvucitabine: Elvucitabine (blinded) 10 mg/day in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
- Lamivudine: Lamivudine (blinded) 300 mg daily in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
- Total: Total of all reporting groups
Arm/Group | Elvucitabine | Lamivudine | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.20) | 36.4 (11.34) | 36.6 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 32 | 29 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 21
  Not Hispanic or Latino | 26 | 29 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: inches] | 68.18 (4.433) | 67.33 (4.325) | 67.77 (4.373)
Weight [Mean (Standard Deviation); unit: pounds] | 162.03 (41.272) | 171.37 (52.582) | 166.58 (47.035)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion Of Participants With Virologic Response For 10 mg/Day Elvucitabine In HIV-1-Infected Participants By 12 Weeks Compared With The Proportion Of Participants With Lamivudine 300 mg/Day
Description: The proportion of participants having achieved a virologic response for elvucitabine 10 mg/day in combination with efavirenz and tenofovir in HIV-1-infected participants over 12 weeks compared with the proportion of participants having achieved a virologic response for lamivudine 300 mg/day in combination with efavirenz and tenofovir. Virologic response was defined as having achieved undetectable (<50 copies/mL) HIV-1 RNA levels from baseline assessment.
Time Frame: 12 weeks
Population: This primary outcome measure used the intent-to-treat population, defined as all randomized participants who took at least 1 dose of study drug and had both a baseline HIV-1 RNA result and at least 1 HIV-1 RNA result after baseline assessment. For this analysis, all participants who discontinued from the study before Week 12 were considered as The Noncompleter=Failure (NC=F).
Measure: Number; unit: percentage of participants
Arm/Group | Elvucitabine | Lamivudine
Number analyzed (Participants) | 37 | 37
percentage of participants
  Week 2 | 13.5 | 8.1
  Week 4 | 16.2 | 10.8
  Week 6 | 27.0 | 35.1
  Week 8 | 35.1 | 54.1
  Week 10 | 54.1 | 56.8
  Week 12 | 56.8 | 70.3
Statistical Analysis 1: Comparison: Elvucitabine vs Lamivudine; The difference in proportions between the group of participants who received lamivudine 300 mg/day (in combination with efavirenz and tenofovir) over 12 weeks and the group of participants who received elvucitabine 10 mg/day (in combination with efavirenz and tenofovir) over 12 weeks along with corresponding 2-sided 95% confidence interval for risk difference using asymptotic normal theory; Test type: Superiority or Other; Risk Difference (RD) = -13.5, 95% CI 2-sided [-35.2 to 8.2]

2. Primary Outcome: The Safety Profile Of Elvucitabine.
Description: Determination of the safety profile of elvucitabine as defined by the frequency, type and severity of treatment-emergent adverse events (AEs) and the frequency of Grade 3 and Grade 4 laboratory abnormalities.
Time Frame: 12 weeks
Population: The analysis population for safety and tolerability was the safety population, defined as all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Elvucitabine, Efavirenz,Tenofovir: Elvucitabine (blinded) 10 mg/day in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
- Lamivudine,Efavirenz,Tenofovir: Lamivudine (blinded) 300 mg daily in combination with open-label efavirenz 600 mg daily and open-label tenofovir 300 mg daily, all administered orally, over 12 weeks. Eligible participants continued with an additional 84 weeks of open-label treatment (through Week 96).
Arm/Group | Elvucitabine, Efavirenz,Tenofovir | Lamivudine,Efavirenz,Tenofovir
Number analyzed (Participants) | 39 | 37
participants
  Treatment emergent adverse events | 36 | 35
  Treatment emergent severe adverse events | 3 | 2
  Treatment related serious adverse events | 0 | 0
  Discontinuations due to adverse events | 2 | 0
  Treatment emergent Grade 3/4 lab abnormalities | 6 | 5

ADVERSE EVENTS:
Time Frame: AE data were collected from enrollment into the study to 96 weeks.
Description: Treatment-emergent AEs are summarized.
Arm/Group | Elvucitabine | Lamivudine
Serious Adverse Events (participants affected / at risk) | 10/39 | 5/37
Other Adverse Events (participants affected / at risk) | 37/39 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elvucitabine (N=39) | Lamivudine (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (3)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Multiple drug overdose intentional (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Elvucitabine (N=39) | Lamivudine (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Auricular swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypogonadism (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Scleral hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Apththous stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (11) | 12 (15)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 3 (3)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (13) | 8 (10)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Painful defaecation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (4)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8) | 7 (8)
Asthenia (General disorders) | 3 (3) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 3 (6)
Feeling drunk (General disorders) | 2 (2) | 0 (0)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (4) | 3 (3)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (5)
Pyrexia (General disorders) | 4 (7) | 8 (13)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (3) | 2 (2)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 6 (9)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Condyloma acuminatum (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (6)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Gonorrhoea (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 3 (3) | 1 (1)
Herpes zoster (Infections and infestations) | 4 (4) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (2)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 2 (5)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (5) | 2 (2)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (3) | 2 (4)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 6 (7)
Staphylococcal infection (Infections and infestations) | 1 (3) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 2 (2)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 11 (14)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0/7 (0) | 1/8 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 2 (3) | 1 (4)
Blood creatine phosphokinase (Investigations) | 1 (3) | 0 (0)
Blood phosphorus decreased (Investigations) | 2 (2) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 2 (4) | 2 (4)
Low density lipoprotein increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0/7 (0) | 1/8 (1)
Tuberculin test positive (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (7)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7) | 6 (8)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 8 (10) | 9 (13)
Headache (Nervous system disorders) | 9 (12) | 7 (10)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 4 (6)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 8 (8)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (6)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Disorientation (Psychiatric disorders) | 2 (2) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6) | 6 (6)
Loss of libido (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Premature ejaculation (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral ulcer (Renal and urinary disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0/7 (0) | 1/8 (2)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast microcalcification (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1/32 (1) | 0/29 (0)
Genital pruritus female (Reproductive system and breast disorders) | 1/7 (1) | 0/8 (0)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1/32 (1) | 0/29 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1/32 (1) | 0/29 (0)
Pruritus genital (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1/7 (2) | 0/8 (0)
Vaginal mucosal blistering (Reproductive system and breast disorders) | 0/7 (0) | 1/8 (1)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (5)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (5)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (7)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug abuser (Social circumstances) | 1 (1) | 0 (0)
Physical abuse (Social circumstances) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting/presenting a manuscript or materials relating to a Study to a publisher, reviewer, or outside person, the Institution shall provide to Sponsor a copy of all such manuscripts or materials, and Sponsor shall have thirty (30) days to review and comment. The Institution shall, upon Sponsor's request, further delay publication or presentation for a period of up to sixty (60) days to allow Sponsor to protect its interests in any Sponsor Inventions.